CLINICAL TRIAL: NCT06222606
Title: Surgery for Thyroid Cancer With or Without Autofluorescence to Prevent Hypoparathyroidism - a Randomized, Controlled Trial
Brief Title: Surgery for Thyroid Cancer With or Without Autofluorescence to Prevent Hypoparathyroidism
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Jacob Kinggaard Lilja-Fischer, MD, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-10-72-120-23
Record Dates: First submitted 2024-01-04; First posted 2024-01-25 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Thyroid Cancer
Keywords: Thyroid Cancer; Surgery; Autofluorescence; Near-Infrared Autofluorescence Imaging; Hypoparathyroidism
MeSH Terms: conditions — Thyroid Neoplasms; Hypoparathyroidism | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: RCT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): Patients randomized to the experimental group will have surgery performed in the exact same manner as in the control group.
- Surgery with EleVision IR camera system (Experimental): In the experimental group, the surgeon will use the EleVision IR camera system (Medtronic, USA) to visualize PGs during surgery. The surgeon will use AF at minimum two timepoints on each side of the neck: First, when the thyroid lobe is exposed and mobilized, and secondly after removal of the thyroid lobe. This is repeated in the contralateral side of the neck in case of TT. If a central neck dissection is performed, the specimen is also examined with AF following removal. Autotransplantation of inadvertently removed PGs may be performed after frozen section histology.
  Interventions: Procedure: Surgery with autofluorescence

INTERVENTIONS:
Procedure: Surgery with autofluorescence — In the experimental group, the surgeon will use the EleVision IR camera system (Medtronic, USA) to visualize parathyroid glands during surgery.
  Arms: Surgery with EleVision IR camera system

SUMMARY:
The study aims to test if use of autofluorescence imaging (AF) reduces the risk of developing hypoparathyroidism (hypoPT) following surgery for thyroid cancer, either total thyroidectomy (TT) or completion hemithyroidectomy (cHT).

DETAILED DESCRIPTION:
Purpose The study aims to test if use of autofluorescence imaging (AF) reduces the risk of developing hypoparathyroidism (hypoPT) following surgery for thyroid cancer, either total thyroidectomy (TT) or completion hemithyroidectomy (cHT).

Background The mainstay of treatment of thyroid cancer is surgery. Many patients will need only surgery with removal of one half of their thyroid gland, a hemithyroidectomy (HT), while others will need to have all of the thyroid gland removed.1 This may be done in one procedure, a total thyroidectomy (TT), or in two procedures with a completion hemithyroidectomy (cHT) after an initial HT. The indication for complete removal of the thyroid gland, may be to remove all cancer tissue, to facilitate adjuvant treatment with radioactive iodine, or both.

Following adequate treatment, overall prognosis is very favorable, with a 3-year overall survival of 98% for all Danish patients diagnosed in 2018.2 Thus, a major point of attention is to minimize treatment-related morbidity, and enable cancer survivorship with as few late-effects as possible.

Surgery for thyroid cancer comes with general surgical risks of bleeding and infection, and specific for thyroid surgery is the risk of injury to nerves to the larynx, which is relatively rare, below 5%. Hypothyroidism is obligatory after TT/cHT, and is seen in 10-15% after HT.

Specific to patients after TT/cHT is damage to the parathyroid glands (PGs), which leads to hypoparathyroidism (hypoPT).

HypoPT is generally thought to be an avoidable surgical complication, but nonetheless it is relatively frequent after surgery for thyroid cancer, depending on the definition applied.3-5 Only patients who have a TT or cHT are at risk of developing hypoPT, since the two contralateral PGs will not have been disturbed and HT is generally not associated with hypoPT.

HypoPT may be transient, but is often permanent. Chronic hypoPT leads to lifelong need for medical surveillance and treatment, and is often difficult to treat. It comes with a risk of health complications (renal and neuropsychiatric), is frequently symptomatic (often cognitive and neuromuscular), and leads to decreased quality of life.6 Thus, there is a need to decrease the risk of hypoPT after surgery for thyroid cancer. Further, due to the favorable prognosis and relatively young age of patients, any improvement will lead to a substantial gain in years lived without complications for each patient, and decreased medical spending for society as a whole. Recently, the national guidelines have been revised to reduce the number of patients who will need TT/cHT and thus be at risk of hypoPT, but still there is a substantial burden of morbidity that needs to be reduced.

Avoidance of hypoPT mainly lies with the surgeon's experience and skills, since identification and preservation of PGs may be very difficult, due to their small size and delicate structure. Identification of PGs is visual, and depends on the surgeon's knowledge of their usual position in relation to the thyroid gland. In the setting of advanced thyroid cancer, preservation of PGs may be extremely difficult, since removal of the primary tumor and metastases adjacent to the PGs is the overwhelming priority.

Recently, it has been discovered that PGs possess unique autofluorescent properties, in that the tissue will return light in a specific wavelength after illumination with infrared light of a specific wavelength. This autofluorescence (AF) may be observed with a hand-held camera system during surgery, allowing the surgeon to more easily visualize and identify PGs.7 This could potentially lead to improved preservation of PGs, and thus decreased risk of hypoPT.

Study design The planned trial is a randomized, controlled superiority trial with two parallel arms. The investigators seek to include patients undergoing surgery for thyroid cancer, who are at risk of developing hypoPT as a complication to surgery. Patients will be randomized 1:1 to surgery with or without the added use of AF during surgery.

Study setting and practical conduct The trial is to be conducted at Aarhus University Hospital, in a collaboration between Department of Otorhinolaryngology - Head & Neck Surgery and Department of Endocrinology. Here, approximately 100 patients undergo surgery for thyroid cancer annually. A further 4-500 patients have thyroid surgery for benign disease, and another approximately 300 patients have surgery for parathyroid disease. Thus, there is a steady high flow of eligible patients, and the hospital as well as the treating surgeons are highly qualified to undertake this study. Autofluorescence imaging with the EleVision IR system is available, and is used ad hoc for thyroid and parathyroid surgery.

Patient flow Patients referred on suspicion of thyroid cancer to the Head and Neck Surgery Clinic at Aarhus University Hospital will be considered for inclusion in the trial. Approximately half of patients with thyroid cancer will need TT or cHT, and will thus be eligible for the trial. The investigators aim to include 110 patients, which should be achievable in approximately two years.

Randomization Following patient consent, an electronic case file will be created in the REDCap electronic data capture tool. Randomization is performed electronically in the dedicated REDCap randomization module.

Randomization will be stratified by TT or cHT.

Intervention Patients randomized to the experimental group will have surgery performed in the exact same manner as in the control group.

In the experimental group, the surgeon will use the EleVision IR camera system (Medtronic, USA) to visualize PGs during surgery. The surgeon will use AF at minimum two timepoints on each side of the neck: First, when the thyroid lobe is exposed and mobilized, and secondly after removal of the thyroid lobe. This is repeated in the contralateral side of the neck in case of TT. If a central neck dissection is performed, the specimen is also examined with AF following removal. Autotransplantation of inadvertently removed PGs may be performed after frozen section histology.

Endpoints HypoPT following surgery is defined as hypocalcemia (ionized plasma calcium levels below lower limit of reference, 1,18 mmol/l), with inappropriately low plasma levels of PTH (assessed by 2 separate measurements) necessitating treatment with active vitamin D, as determined by the treating physician.

Deviation from standard treatment All patients, whether randomized to standard or experimental treatment arm, will receive treatment according to national clinical guidelines published by the Danish Thyroid Cancer Group (DATHYRCA).1 The extent of surgery will be exactly the same in either group, and will not deviate from standard treatment.

Sample size The investigators estimate that the rate of hypoPT requiring medical treatment in the control group will be approximately 30%. A reduction to 10% will be clinically significant, and statistically significant at α=0.05 with a power of β=0.8 with inclusion of 98 patients. To allow for dropouts, the investigators aim to include 110 patients, which should be achievable in approximately two years.

Interim analysis The investigators plan to perform an interim analysis after inclusion of 50 patients with available data on the primary endpoint. The trial may be terminated if the investigators are able to show that it would be highly unlikely to reach the primary endpoint. This may be due to no effect of the intervention, or a lower than expected risk of hypoPT in the control group. Both scenarios would make it highly unlikely to reach the primary endpoint of the study.

Statistical analysis plan For the primary endpoint, relative risk for hypoPT will be calculated along with its associated 95% confidence interval, and a p-value will be calculated from a chi2-test. The investigators will provide a crude estimate, as well as adjusted for operating surgeon, or suspicion of lymph node metastases on imaging and/or planned neck dissection.

For secondary endpoints, a similar analysis will be performed for categorical data (Permanent hypoPT; extent of surgery; complications). Continuous data (ioPTH reduction, time to resolution of hypoPT, number of days hospitalized) will be described and analysed using a t-test, or ranksum test in case of non-normal data. Survival endpoints will be described by a hazard ratio with 95% confidence interval.

Patient characteristics, including demographics, disease status and treatment will be characterized using descriptive statistics only.

Risk, side effects and disadvantages Use of AF during surgery involves nothing but 2 to 5 minutes of illumination of the surgical field with infrared light through a hand-held camera, which displays an image on a monitor in which the infrared wavelengths are converted to wavelengths visual to the human eye. The potential effect of use of AF in thyroid cancer surgery is to make the surgeon more aware of the PGs, and thus incite the surgeon to change his/her strategy in a more patient-safe direction.

Illumination of the surgical field with infrared light has no biological effect, cannot be felt, and poses no danger to the patient. Thus, the intervention should not lead to discomfort or pain, has no known side effects and would not pose a risk to the patient.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years and able to give informed consent.
* Suspicion or diagnosis of thyroid cancer.
* Planned total thyroidectomy or completion thyroidectomy.
* Normocalcemia prior to surgery.

Exclusion Criteria:

* Planned simultaneous parathyroid surgery.
* Treatment with active vitamin D analogues.
* eGFR < 30.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Hypoparathyroidism | 6 and 12 months
  Proportion of patients who develop transient or permanent hypoPT requiring medical treatment with active vitamin D. HypoPT is diagnosed and treated according to protocol.

SECONDARY OUTCOMES:
Permanent hypoparathyroidism | 6 and 12 months
  Proportion of patients who develop permanent hypoPT.
Intra-operative reduction in plasma concentration of PTH. | During surgery
  PTH is measured before start and immediately after surgery.
Time to resolution of transient hypoPT. | 12 months
  Time to resolution of transient hypoPT.
Number of days hospitalized | 30 days
  Number of days hospitalized during first 30 days after surgery.
Oncological and composite outcomes | 2 years
  Overall survival. Disease-free survival. Disease- and hypoPT-free survival.

OTHER OUTCOMES:
Histology report | 1 week
  Number of parathyroid glands (PGs) and lymph node metastases identified.
Extent of surgery | During surgery
  Central neck dissection, lateral neck dissection, autotransplantation of PGs.
Complications | 30 days
  Bleeding, infection, recurrent nerve palsy, serious adverse events.
AF pattern | During surgery
  Description of AF pattern of tissue during central neck dissection / exploration, specifically with regards to lymph nodes, lymph node metastases and PGs.
Parathyroid gland identification | During surgery
  Surgeons assessment of identified parathyroid glands with or without autofluorescence.

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Pseudonymized IPD may be shared for meta-analysis, if IRB approval is granted.